CLINICAL TRIAL: NCT04461756
Title: A Phase I Exploratory Study to Assess the Pharmacokinetics of Single Inhaled Dose of Cannabis (Delta-9-Tetrahydrocannabinol / Cannabidiol) Administered by Vaporization Using a 4-Day Dose Titration In Healthy Male And Female Volunteers
Brief Title: Safety and Pharmacokinetics of Vaped Cannabis in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetra Bio-Pharma (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPP001-Ph1-03
Record Dates: First submitted 2020-03-10; First posted 2020-07-08 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volonteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inhaled THC/CBD (PPP001) (Experimental)
  Interventions: Drug: PPP001

INTERVENTIONS:
Drug: PPP001 — inhalation (vape)

SUMMARY:
The primary objective of this study was to evaluate the pharmacokinetics (PK) of THC, 11-OH-THC and CBD following a single inhaled dose of PPP001 administered by vaporization.

The secondary objective of this study was to determine the safety and tolerability of THC and CBD after a single inhaled dose of PPP001 administered by vaporization in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within 21.0 to 32.0 kg/m2, inclusively
* A light-, non- or ex-smoker of nicotine
* A history of recreational cannabis use (at least 10 times in the last 5 years)
* Consumed cannabis in the last 3 months before Day 1 of the study, but not within 1 month before Day 1 of the study
* Presence of intact oral mucosa
* Able to follow instructions at the training vaporizing session
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must have been without clinical significance, as determined by an investigator
* No clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs), or ECG, as determined by an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events [Safety and Tolerability] | over 5 days
  To evaluate treatment-related adverse events of PPP001
Biochemistry test results [Safety and Tolerability] | over 5 days
  Number of subjects with alkaline phosphatase and alanine aminotransferase (ALT) increase
Temperature [Safety and Tolerability] | over 5 days
  Oral temperature in Celsius
Pulse rate [Safety and Tolerability] | over 5 days
  Pulse rate (in beats per minute)
Blood pressure [Safety and Tolerability] | over 5 days
  Blood pressure (systolic/diastolic blood pressure in mm Hg)
Clinically significant ECG abnormalities [Safety and Tolerability] | over 5 days
  Number of subjects with clinically significant ECG abnormalities (measured with a 12-lead ECG)
Plasma concentrations of delta-9-tetrahydrocannabinol produced by PPP001 were determined. (pharmacokinetics) | over 5 days
Plasma concentrations of 11-OH-delta-9-tetrahydrocannabinol produced by PPP001 were determined. (pharmacokinetics) | over 5 days
Plasma concentrations of cannabidiol produced by PPP001 were determined. (pharmacokinetics) | over 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alta sciences, Montreal, Quebec, Canada